CLINICAL TRIAL: NCT00060827
Title: Head Impact Recording Technology for Field Applications
Brief Title: Measuring Head Impacts in Sports
Status: Withdrawn | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Other Study IDs: R44HD040743-02 (NIH)
Record Dates: First submitted 2003-05-14; First posted 2003-05-15 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2004-03

CONDITIONS: Brain Injuries; Brain Concussion
Keywords: Mild traumatic brain injury
MeSH Terms: conditions — Brain Injuries; Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Head Impact Recording Technology (HIRT)

SUMMARY:
Head impacts in sports can lead to brain injury even when the participant is wearing a helmet. The forces that contribute to brain injury from sports-related head impacts are not well understood. This study will test a new device to measure the speed of head impacts among football players.

DETAILED DESCRIPTION:
Each year, 50 to 70 million people in the United States participate in helmeted and unhelmeted sports with the potential for head impacts. Such sports include football, soccer, hockey, basketball, and boxing. Participating in these sports carries the risk of mild traumatic brain injury (MTBI). The biomechanics of head impacts that result in concussions or other MTBIs are not well understood; however, it is thought that such impacts correlate with head accelerations. Currently, there is no system that allows researchers to measure head acceleration in a large number of individuals during actual play. This is a major obstacle in understanding the mechanism of MTBI and its prevention. This study will evaluate a newly designed miniature device that uses Head Impact Recording Technology (HIRT) to quantify head acceleration during impact in actual sports play.

One hundred college football players will be enrolled in the study. Data from HIRT-instrumented helmets will be collected during normal team practice and games throughout a 5-month football season. Data collected will be assessed to determine the incidence, magnitude, and duration of head acceleration during impacts on the sports field.

ELIGIBILITY:
Inclusion Criteria

* College football players

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Impact Severity | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Rick Greenwald, Ph.D., Principal Investigator
Locations (1):
- Penn State University, State College, Pennsylvania, United States